CLINICAL TRIAL: NCT07142798
Title: Efficacy of Bismuth/Amoxicillin/Potassium-competitive Acid Blocker Triple Therapy for the Treatment of Helicobacter Pylori Infection in Taiwan
Brief Title: to Assess the Eradication Rate of 14-day Bismuth/Amoxicillin/PCAB Triple Therapy for the Treatment of Helicobacter Pylori Infection
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Collaborators: An-Nan Hospital, China Medical University (Other)
Responsible Party: Principal Investigator, DENG-CHYANG WU, Professor, Kaohsiung Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20240204
Record Dates: First submitted 2025-08-19; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: HELICOBACTER PYLORI INFECTIONS
Keywords: Helicobacter pylori therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Helicbpacyer pylori infection (Experimental): Helicbpacyer pylori infection
  Interventions: Drug: Bismuth amoxilillin potassium

INTERVENTIONS:
Drug: Bismuth amoxilillin potassium — vonoprazan 20mg， Twice a day amoxicillin 750mg，Four times a day tripotassium dicitrate bismuthate 300mg，Four times a day for 14 days

SUMMARY:
To assess the efficacy and safety of 14-day bismuth/amoxicillin/PCAB triple therapy for the treatment of Helicobacter pylori infection in Taiwan

ELIGIBILITY:
Inclusion Criteria:

Subjects infected with Helicobacter pylori.

Exclusion Criteria:

1. Those who are allergic to the drugs used in this research.
2. Those who have had stomach surgery.
3. Those with severe liver cirrhosis or uremia or malignant tumors.
4. Women who are pregnant or breastfeeding. If you have drug allergies or pregnant women or breast-feeding women during the test period, you can withdraw from the test early.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Eradicaton rate of Helicobacter pylori | 6 weeks after finishing study drugs
  13CUBT

SECONDARY OUTCOMES:
evaluate side effect | 2days after taking medicine
  evaluate drugy side effect by Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No